CLINICAL TRIAL: NCT04591197
Title: Flumatinib Efficacy and Safety for New Diagnosed Chronic Phase Chronic Myeloid Leukemia : A Prospective, Multi-center, Single Arm Study
Brief Title: Flumatinib Efficacy and Safety for New Diagnosed Chronic Phase Chronic Myeloid Leukemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, xuna, Associate chief physician, Nanfang Hospital, Southern Medical University
Other Study IDs: HS-NF-2020
Record Dates: First submitted 2020-10-15; First posted 2020-10-19 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Validity and Safety

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall survival (OS)of Chronic myeloid leukemia (CML) has been significantly improved since the advent of Tyrosine kinase inhibitors (TKIs) .Nevertheless, there still exists a amount of patients who has poor response or intolerance for TKI drugs( Imatinib, dasatinib, nilotinib). Flumatinib has been shown to be a more potent inhibitor of BCR-ABL1 tyrosine kinase than imatinib,and it aslo has better security when compared to other TKIs(Imatinib, dasatinib, nilotinib).It will be a better chioce for CML patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, both male and female;
2. New Diagnosed Chronic Phase Chronic Myeloid Leukemia.
3. Within half a year after diagnosis of CML;
4. Previous TKIs treatment was less than 2 weeks;
5. The pregnant test of female patients was negative (within 7 days before medication before enrollment);
6. Informed consent of the patient or his legal representative

Exclusion Criteria:

1. T315I mutation is known to exist;
2. Rare atypical transcript types that cannot be standardized internationally;
3. Received TKI drugs for more than 2 weeks before enrollment;
4. Received interferon therapy for more than 3 months before enrollment;
5. Received other anti-CML drugs (except hydroxyurea) for more than 2 weeks or surgical treatment (including hematopoietic stem cell transplantation)
6. patients who participate in other clinical studies at the same time;
7. patients who having had major surgery or not recovered from surgery within 4 weeks;
8. patients who having history of malignant tumor
9. Woman who is pregnant or nursing
10. Eastern Cooperative Oncology Group Physical Performance Status Score (ECOG PS) > 3;
11. Patients known to be allergic or contraindicated to the study drug (APIs and/or excipients).
12. A clear history of neurological or psychiatric disorders, including epilepsy or dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: New diagnosed CML-CP patients who are more than 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-12-09 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
MMR rates at 12 months | 12 monts
  MMR(BCR/ABL(IS)<0.1%) at 12 months after treating

SECONDARY OUTCOMES:
VEMR rates at 4 weeks | 4 weeks
  VEMR((BCR-ABL1/ABL1≤ 40% on the International Scale) at 4weeks after treating

CONTACTS AND LOCATIONS:
Locations (1):
- NanfangH, Guangzhou, Guangdong, China